CLINICAL TRIAL: NCT00163189
Title: Evolution Of Growth Rate In Children With Growth Retardation Related To Long-term Corticotherapy And Treated By Genotonorm
Brief Title: Evolution Of Growth Rate In Children With Growth Retardation Due to Glucocorticosteroid Therapy And Treated By Genotonorm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6281271; 2004-002992-17 (EudraCT Number)
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2015-06

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somatropin (Experimental)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Liquid, daily, during 3 years and extended to 5 years Dosage: 0,46 mg/kg/week - the maximum dose should not exceed 50 µg/kg/day

SUMMARY:
To estimate the evolution of height and growth rate over 5 years of growth hormone (GH) treatment To estimate the prognostic factors of growth rate with GH treatment To confirm the good clinical and biological safety of GH treatment in such children

ELIGIBILITY:
Inclusion Criteria:

* Glucocorticosteroid treatment for 12 months at least
* Bone age < 15 years for a boy and < 13 years for a girl
* Child measured height < - 2 SD, Child currently treated by GH

Exclusion Criteria:

* Known diabetes (type 1 or type 2)
* A previous history of intolerance or hypersensitivity to the study drug or to drugs with similar chemical structures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- France (19):
  - Hôpital Nord, Amiens
  - Centre Hospitalier Intercommunal d'Annemasse-Bonneville, Service de Pédiatrie et Néonatologie, Annemasse
  - Hôpital Saint Jacques, Besançon
  - Groupe hospitalier Est- Hôpital Femme, Mère, Enfant, Bron
  - Groupe hospitalier Est-Hôpital Femme, Mère, Enfant, Bron
  - CHU d'Estaing, Clermont-Ferrand
  - CHU de Grenoble, Hôpital Couple enfant., Grenoble
  - CHU Timone Enfants, Marseille
  - Hôpital Arnaud De Villeneuve, Montpellier
  - CHU de Nantes, Hôpital Mère Enfant, Nantes
  - Hôpital Lenval, Nice
  - Hôpital Robert Debré, Paris
  - Hôpital Armand Trousseau, Paris
  - Groupe Hospitalier Necker - Enfants Malades, Paris
  - Centre de Perharidy, Roscoff
  - CHU Charles Nicolle, Rouen
  - Service de Pédiatrie- Centre Hospitalier Intercommunal, Saint-Germain-en-Laye
  - Hôpital des Enfants, Toulouse
  - CHU Tours - Centre Pediatrique Gatien de Cocheville, Tours

REFERENCES:
- [Derived] Basmaison O, Ranchin B, Zouater H, Robertson A, Gomez R, Koppiker N. Efficacy and safety of recombinant growth hormone treatment in children with growth retardation related to long-term glucocorticosteroid therapy. Ann Endocrinol (Paris). 2019 Sep;80(4):202-210. doi: 10.1016/j.ando.2019.02.001. Epub 2019 Mar 4. PMID 30910221
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281271&StudyName=Evolution%20Of%20Growth%20Rate%20In%20Children%20With%20Growth%20Retardation%20due%20to%20Glucocorticosteroid%20Therapy%20And%20Treated%20By%20Genotonorm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reason 'Study Terminated by Sponsor' mentioned in the participant flow indicates the termination of study at a site (due to Good Clinical Practice [GCP] compliance issues) and does not reflect the overall status of study.
Groups:
- Genotonorm: Genotonorm 0.46 milligram per kilogram (mg/kg) administered weekly, divided into 7 daily subcutaneous injections (maximum dose not exceeding 50 microgram [mcg]/kg/day) for up to 60 months.
Period: Overall Study
Arm/Group | Genotonorm
Started | 98
Completed | 35
Not Completed | 63
Not completed — Other | 6
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — Death | 3
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 7
Not completed — Study terminated by sponsor | 11
Not completed — Withdrawal by Subject | 11
Not completed — Did not meet continuation criterion | 16

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants (including a site with GCP issues) who had received at least 1 study dose of growth hormone (GH).
Arm/Group | Genotonorm
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 74

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) for Chronological Age (CA) at Month 36: Full Analysis Population
Description: Height was measured using a wall mounted device (example, Harpenden stadiometer). The standing height of the participant was measured two times and the mean of these measurements was recorded. Height SDS CA Yx = (height Yx - reference mean for CA Yx) / reference SD for CA Yx; Yx refers to the value at particular timepoint x. Height in SDS was calculated using Sempe reference means and SD for height. CA calculated as integer (Date of height measurement-Date of birth)/365.25*12.
Time Frame: Baseline, Month 36
Population: Full analysis set (FAS) included all participants (excluding a site with GCP issues) who had received at least 1 injection of GH and had at least 1 post-Baseline measurement of height. Here "n" signifies those participants who were evaluable for the specified time point.
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
Standard Deviation Score (SDS)
  Baseline (n=58) | -2.91 (1.19)
  Change at Month 36 (n=30) | 0.80 (1.03)
Statistical Analysis 1: Comparison: Genotonorm; Month 36; Test type: Superiority or Other; p < 0.001, Student's paired t-test

2. Primary Outcome: Change From Baseline in Height Standard Deviation Score (SD) for Chronological Age (CA) at Month 36: Per Protocol (PP) Population
Description: as for outcome 1
Time Frame: Baseline, Month 36
Population: PP analysis set included all participants (excluding a site with GCP issues) who received at least 1 dose of GH, had at least 1 subsequent rating of height, no major protocol violation till first 3 years post initiation of treatment and total GH treatment duration of 36 months or more. "n"=participants evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 21
SDS
  Baseline (n=21) | -2.86 (0.89)
  Change at Month 36 (n=19) | 0.81 (1.18)
Statistical Analysis 1: Comparison: Genotonorm; Month 36; Test type: Superiority or Other; p = 0.008, Student's paired t-test

3. Secondary Outcome: Mean Height
Description: The standing height measurements were performed using a wall mounted device (example Harpenden Stadiometer). The standing height of the participant was measured two times and the mean of these measurements was recorded.
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: FAS included all participants (excluding a site with GCP issues) who had received at least 1 injection of GH and had at least 1 post-Baseline measurement of height. Here "n" signifies those participants who were evaluable for the specified time point.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
centimeters (cm)
  Baseline (n=58) | 133.9 (15.7)
  Month 12 (n=50) | 139.5 (16.8)
  Month 24 (n=41) | 146.0 (16.4)
  Month 36 (n=30) | 150.4 (16.0)
  Month 48 (n=14) | 152.4 (16.0)
  Month 60 (n=9) | 156.0 (11.3)

4. Secondary Outcome: Mean Height Standard Deviation Score (SDS) for Bone Age (BA)
Description: The standing height measurements were performed using a wall mounted device (example Harpenden Stadiometer). The standing height of the participant was measured two times and the mean of these measurements was recorded. Height SDS BA Yx = (height Yx - reference mean for BA Yx) / reference SD for BA Yx; Yx refers to the value at particular timepoint x. Height in SDS was calculated using Sempe reference means and SD for height. BA was estimated locally using an X-ray from the left wrist and hand.
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
SDS
  Baseline (n=51) | -0.29 (1.15)
  Month 12 (n=40) | -0.36 (1.52)
  Month 24 (n=29) | 0.11 (1.36)
  Month 36 (n=24) | 0.14 (1.48)
  Month 48 (n=13) | -0.26 (1.28)
  Month 60 (n=7) | -0.19 (1.15)

5. Secondary Outcome: Annual Growth Rate (AGR)
Description: AGR at Yx was derived by subtracting AGR at baseline from Yx value. AGR was calculated each year and re scaled to 1 year if the interval between Yx and Y[x-1] was not 365 days, as long as a participant remained in the study. AGR at Yx was calculated using the previous height measurements (Y[x-1]) and height recorded at Yx (AGR Yx = [height Yx-height Y{x-1}] / ([date of Yx - date of Y{x-1}] /365.25). Yx refers to the value at particular timepoint x.
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
cm/year
  Baseline (n=52) | 3.0 (2.0)
  Month 12 (n=49) | 6.7 (2.6)
  Month 24 (n=41) | 6.0 (2.7)
  Month 36 (n=30) | 5.9 (2.7)
  Month 48 (n=14) | 4.8 (2.5)
  Month 60 (n=9) | 4.9 (3.0)

6. Secondary Outcome: Growth Rate (GR) Standard Deviation Score (SDS) for Bone Age (BA)
Description: GR SDS BA Yx = (GR Yx - reference mean for BA Yx) / reference SD for BA Yx; Yx refers to the value at particular timepoint x. GR in SDS was calculated using Sempe reference means and SD for GR. BA was estimated locally using an X-ray from the left wrist and hand.
Time Frame: Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
SDS
  Month 12 (n=36) | -0.13 (2.15)
  Month 24 (n=25) | 0.07 (2.51)
  Month 36 (n=20) | 0.05 (1.94)
  Month 48 (n=11) | -1.00 (1.38)
  Month 60 (n=7) | -0.43 (1.22)

7. Secondary Outcome: Growth Rate (GR) Standard Deviation Score (SDS) for Chronological Age (CA)
Description: GR SDS CA Yx = (GR Yx - reference mean for CA Yx) / reference SD for CA Yx; Yx refers to the value at particular timepoint x. GR in SDS was calculated using Sempe reference means and SD for GR. CA calculated as integer (Date of height measurement-Date of birth)/365.25*12.
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
SDS
  Baseline (n=52) | -2.04 (2.03)
  Month 12 (n=49) | 1.77 (4.29)
  Month 24 (n=41) | 5.26 (16.79)
  Month 36 (n=29) | 3.64 (9.06)
  Month 48 (n=13) | 0.93 (2.73)
  Month 60 (n=9) | 1.40 (1.71)

8. Secondary Outcome: Body Mass Index (BMI)
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2).
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
kg/m^2
  Baseline (n=58) | 19.4 (3.6)
  Month 12 (n=50) | 19.1 (3.1)
  Month 24 (n=41) | 19.4 (3.0)
  Month 36 (n=30) | 19.4 (2.4)
  Month 48 (n=14) | 19.7 (3.0)
  Month 60 (n=9) | 20.8 (3.3)

9. Secondary Outcome: Change From Baseline in Height at Month 12, 24, 36, 48 and 60
Description: as for outcome 3
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
cm
  Baseline (n=58) | 133.9 (15.7)
  Change at Month 12 (n=50) | 6.8 (2.8)
  Change at Month 24 (n=41) | 12.9 (4.7)
  Change at Month 36 (n=30) | 18.8 (6.1)
  Change at Month 48 (n=14) | 23.9 (8.5)
  Change at Month 60 (n=9) | 30.3 (7.6)

10. Secondary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) for Chronological Age (CA) at Month 12, 24, 48 and 60
Description: The standing height measurements were performed using a wall mounted device (example Harpenden Stadiometer). The standing height of the participant was measured two times and the mean of these measurements was recorded. Height SDS CA Yx = (height Yx - reference mean for CA Yx) / reference SD for CA Yx; Yx refers to the value at particular timepoint x. Height in SDS was calculated using Sempe reference means and SD for height. CA calculated as integer (Date of height measurement-Date of birth)/365.25*12.
Time Frame: Baseline, Month 12, 24, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
SDS
  Baseline (n=58) | -2.91 (1.19)
  Change at Month 12 (n=50) | 0.28 (0.57)
  Change at Month 24 (n=41) | 0.57 (0.95)
  Change at Month 48 (n=14) | 0.82 (1.42)
  Change at Month 60 (n=9) | 0.75 (1.13)

11. Secondary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) for Bone Age (BA) at Month 12, 24, 36, 48 and 60
Description: as for outcome 4
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
SDS
  Baseline (n=51) | -0.29 (1.15)
  Change at Month 12 (n=36) | -0.02 (0.99)
  Change at Month 24 (n=26) | 0.28 (1.18)
  Change at Month 36 (n=21) | 0.31 (1.17)
  Change at Month 48 (n=13) | -0.08 (1.30)
  Change at Month 60 (n=7) | 0.01 (1.33)

12. Secondary Outcome: Change From Baseline in Bone Age (BA) at Month 12, 24, 36, 48 and 60
Description: BA was estimated locally using an X-ray from the left wrist and hand.
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
months
  Baseline (n=58) | 117.9 (34.6)
  Change at Month 12 (n=37) | 17.8 (11.0)
  Change at Month 24 (n=32) | 28.2 (17.9)
  Change at Month 36 (n=23) | 36.5 (17.8)
  Change at Month 48 (n=13) | 52.8 (21.2)
  Change at Month 60 (n=7) | 70.0 (27.0)

13. Secondary Outcome: Ratio of Bone Age (BA) to Chronological Age (CA)
Description: BA was estimated locally using an X-ray from the left wrist and hand. CA at the date of corresponding X-ray (Date of X-ray - Date of birth)/365.25. Ratio of BA/CA at each annual study visit was calculated.
Time Frame: Baseline, Month 12, 24, 36, 48, 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Genotonorm
Number analyzed (Participants) | 58
ratio
  Baseline (n=58) | 0.78 (0.10)
  Month 12 (n=37) | 0.82 (0.11)
  Month 24 (n=32) | 0.80 (0.09)
  Month 36 (n=23) | 0.79 (0.10)
  Month 48 (n=13) | 0.81 (0.08)
  Month 60 (n=7) | 0.85 (0.10)

14. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs include both SAEs and non-SAEs.
Time Frame: Baseline up to 28 days after last study treatment
Population: Safety analysis set included all participants (including a site with GCP issues) who had received at least 1 study dose of GH.
Measure: Number; unit: participants
Arm/Group | Genotonorm
Number analyzed (Participants) | 98
participants
  AEs | 84
  SAEs | 45

15. Other Pre Specified Outcome: Number of Participants With Significant Changes in Physical Examinations
Description: Number of participants with clinically significant physical examinations changes since previous visit were reported. Physical examination including estimation of pubertal stage and blood pressure measurement;
Time Frame: Baseline, Month 12, 24, 36, 48, 60, End of Treatment (EOT)
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Genotonorm
Number analyzed (Participants) | 98
participants
  Baseline (n=93) | 1
  Month 12 (n=93) | 16
  Month 24 (n=72) | 16
  Month 36 (n=52) | 5
  Month 48 (n=23) | 4
  Month 60 (n=12) | 2
  EOT (n=44) | 11

16. Other Pre Specified Outcome: Number of Participants With at Least 1 Medical or Surgical History
Time Frame: Screening
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Genotonorm
Number analyzed (Participants) | 98
participants | 67

17. Other Pre Specified Outcome: Number of Participants Who Received Concomitant Medications
Time Frame: Baseline up to Month 60
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Genotonorm
Number analyzed (Participants) | 98
participants | 98

18. Other Pre Specified Outcome: Fasting Serum Insulin Like Growth Factor-1 (IGF-1) Levels
Time Frame: Screening, Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Genotonorm
Number analyzed (Participants) | 98
nanogram per milliliter (ng/mL)
  Screening (n=93) | 335 (157)
  Month 6 (n=63) | 604 (291)
  Month 12 (n=71) | 538 (268)
  Month 18 (n=47) | 624 (251)
  Month 24 (n=62) | 579 (262)
  Month 30 (n=50) | 559 (250)
  Month 36 (n=44) | 511 (186)
  Month 42 (n=22) | 555 (224)
  Month 48 (n=21) | 581 (244)
  Month 54 (n=16) | 593 (184)
  Month 60 (n=10) | 501 (180)

19. Other Pre Specified Outcome: Fasting and Postprandial Plasma Glucose Levels at Month 12, 24, 36, 48 and 60
Description: Fasting and 2 hours plasma glucose levels were assessed using standard oral glucose tolerance test (OGTT).
Time Frame: Screening, Month 12, 24, 36, 48, 60
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milli mole per liter (mmol/L)
Arm/Group | Genotonorm
Number analyzed (Participants) | 98
milli mole per liter (mmol/L)
  Glucose Fasting: Screening (n=91) | 4.5 (0.7)
  Glucose Fasting: Month 12 (n=69) | 4.6 (0.7)
  Glucose Fasting: Month 24 (n=59) | 4.7 (0.6)
  Glucose Fasting: Month 36 (n=45) | 4.6 (0.5)
  Glucose Fasting: Month 48 (n=20) | 4.7 (0.4)
  Glucose Fasting: Month 60 (n=14) | 4.5 (0.6)
  Glucose Postprandial: Screening (n=94) | 5.6 (1.2)
  Glucose Postprandial: Month 12 (n=66) | 6.1 (1.4)
  Glucose Postprandial: Month 24 (n=59) | 6.1 (1.4)
  Glucose Postprandial: Month 36 (n=41) | 6.4 (1.6)
  Glucose Postprandial: Month 48 (n=19) | 6.1 (1.1)
  Glucose Postprandial: Month 60 (n=13) | 6.3 (1.5)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Genotonorm
Serious Adverse Events (participants affected / at risk) | 45/98
Other Adverse Events (participants affected / at risk) | 81/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotonorm (N=98)
Gastroenteritis (Infections and infestations) | 8
Sepsis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Varicella (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Empedobacter brevis infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Gastroenteritis cryptosporidial (Infections and infestations) | 1
Gastroenteritis rotavirus (Infections and infestations) | 1
Nail bed infection (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Nephrotic syndrome (Renal and urinary disorders) | 7
Renal failure (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 1
Rectal stenosis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Varices oesophageal (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Headache (Nervous system disorders) | 2
Benign intracranial hypertension (Nervous system disorders) | 1
Cerebral venous thrombosis (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Syncope vasovagal (Nervous system disorders) | 1
Abdominal injury (Injury, poisoning and procedural complications) | 1
Accident (Injury, poisoning and procedural complications) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Cataract operation (Surgical and medical procedures) | 1
Gastrostomy closure (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Thoracic operation (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Cataract (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Hypovolaemic shock (Vascular disorders) | 2
Intermittent claudication (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Subvalvular aortic stenosis (Cardiac disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Depression (Psychiatric disorders) | 2
Cytolytic hepatitis (Hepatobiliary disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Polycystic ovaries (Reproductive system and breast disorders) | 1
Treatment noncompliance (Social circumstances) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotonorm (N=98)
Bronchitis (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 6
Tonsillitis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 5
Influenza (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 4
Varicella (Infections and infestations) | 4
Ear infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Otitis media (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Chikungunya virus infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Dermatophytosis (Infections and infestations) | 1
Eye infection toxoplasmal (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Penile infection (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Trichophytosis (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Duodenitis (Gastrointestinal disorders) | 2
Gingivitis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Odynophagia (Gastrointestinal disorders) | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1
Gingival hypertrophy (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Scoliosis (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Knee deformity (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 3
Skin striae (Skin and subcutaneous tissue disorders) | 3
Dermatomyositis (Skin and subcutaneous tissue disorders) | 2
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Scar (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Asthenia (General disorders) | 8
Pyrexia (General disorders) | 7
Fatigue (General disorders) | 2
Chest pain (General disorders) | 1
Injection site pain (General disorders) | 1
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Cataract (Eye disorders) | 4
Conjunctivitis (Eye disorders) | 3
Ocular hypertension (Eye disorders) | 3
Papilloedema (Eye disorders) | 2
Uveitis (Eye disorders) | 2
Chalazion (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Myopia (Eye disorders) | 1
Night blindness (Eye disorders) | 1
Periorbital disorder (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Vitritis (Eye disorders) | 1
Insulin-like growth factor increased (Investigations) | 13
Weight decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 11
Dysuria (Renal and urinary disorders) | 2
Enuresis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 1
Hemicephalalgia (Nervous system disorders) | 1
Hyperreflexia (Nervous system disorders) | 1
Hypotonia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Haemolysis (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypertension (Vascular disorders) | 4
Thrombosis (Vascular disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Otorrhoea (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Hypertrophic cardiomyopathy (Cardiac disorders) | 1
Cushingoid (Endocrine disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Vasculitis (Immune system disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 2
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 1
Hospitalisation (Surgical and medical procedures) | 1
Pityriasis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.